CLINICAL TRIAL: NCT07019701
Title: Gas Composition in the Hypopharynx During High-flow Oxygen Therapy Through Nasal Cannula or Face Mask, or During Standard Oxygen Therapy Through a Non-Rebreather Face Mask in Healthy Volunteers
Brief Title: Gas Composition in the Hypopharynx During High-flow or Standard Oxygen Therapy Through Face Mask in Healthy Volunteers
Acronym: O2-OXIMETRY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HFNC2-OXIMETRY
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers; HFNC; high flow oxygen; oximetry; capnometry; hypopharynx; standard oxygen therapy; oxygen face mask
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxygen therapy (Experimental): High flow oxygen through nasal cannula and face mask and standard oxygen therapy through non-rebreather face mask, and measurement of oxygen and carbon dioxide fraction in the hypopharynx High flow oxygen through nasal cannula and face mask, and standard oxygen therapy through non-rebreather face mask, and measurement of oxygen and carbon dioxide fraction in the hypopharynx of healthy volunteers in different physiological conditions
  Interventions: Device: High flow oxygen through nasal cannula and face mask and standard oxygen therapy through non-rebreather face mask, and measurement of oxygen and carbon dioxide fraction in the hypopharynx

INTERVENTIONS:
Device: High flow oxygen through nasal cannula and face mask and standard oxygen therapy through non-rebreather face mask, and measurement of oxygen and carbon dioxide fraction in the hypopharynx — High flow oxygen through nasal cannula and face mask, and standard oxygen therapy through non-rebreather face mask, and measurement of oxygen and carbon dioxide fraction in the hypopharynx of healthy volunteers in different physiological conditions

SUMMARY:
The COVID-19 pandemic has become a huge global problem, affecting all spheres of human life, resulting in enormous social, economic consequences and human tragedies. With very decent results of treatment of patients of average severity in the conditions of bed units, the results of treatment of the most severe category - patients of intensive care units who required tracheal intubation remain extremely unsatisfactory. According to different data, mortality in this category of patients reaches 80-90%. However, observational, randomized studies and their meta-analyses have shown high efficiency of high-flow oxygen therapy through nasal cannulas, reaching 50-60%. Some pilot bench studies (on manikins) have shown the advantages of high-flow oxygen therapy over standard oxygen therapy in reducing anatomical dead space and preserving a given inspiratory fraction of oxygen in the laryngeal pharynx of the manikin, but the actual state of the laryngeal pharyngeal gas composition was not studied. Some patients breathe through open mouth that decreases the efficacy oh high flow oxygen through nasal cannula. The aim of the study is to measure the inspiratory (FiO2) and expiratory (FeO2) oxygen fractions and the inspiratory and expiratory carbon dioxide fractions (FiCO2 and FeCO2, respectively) in the hypopharynx of healthy volunteers during high-flow oxygen therapy through nasal cannula and face mask, and during standard oxygen therapy through non-rebreather face mask under different physiological conditions.

DETAILED DESCRIPTION:
Randomized controlled trials showed reduction of tracheal intubation in high- flow oxygen therapy through nasal cannula group in patients with acute respiratory failure as compared to standard oxygen therapy and noninvasive ventilation before Coronavirus disease-19 (COVID-19) pandemic.

The World Health Organization (WHO) declared the outbreak a pandemic of COVID-19 on March 11th, 2020. Since then observational, randomized studies and their meta-analyses have shown the high effectiveness of high-flow oxygen therapy through nasal cannulas (HFNC), reaching 50-60% in acute hypoxemic respiratory failure.

Bench studies showed the advantages of HFNC compared with standard oxygen therapy, consisting in reducing the anatomical dead space and maintaining a given inspiratory oxygen fraction in the hypopharynx of the mannequin, but the actual state of the gas composition of the hypopharynx during HFNC was not studied. Some patients breathe through open mouth that decreases the efficacy oh high flow oxygen through nasal cannula.

The aim of the study is to measure the inspiratory (FiO2) and expiratory (FeO2) oxygen fractions and the inspiratory and expiratory carbon dioxide fractions (FiCO2 and FeCO2, respectively) in the hypopharynx of healthy volunteers during high-flow oxygen therapy through nasal cannula and face mask, and during standard oxygen therapy through non-rebreather face mask under different physiological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Age 18-50 years
* Written informed consent.

Exclusion Criteria:

* Any primary or secondary lung diseases (COPD, bronchial asthma, interstitial lung diseases, metastatic lung disease, lung cancer)
* Any chronic diseases that can cause respiratory disorders (chronic heart failure, liver cirrhosis, systemic connective tissue diseases, cancer, neuromuscular diseases etc)
* Heart rhythm disturbances
* Body mass index more than 30 kg/m2
* Swallowing disorders
* History of epileptic syndrome
* Recent head surgery or anatomy that precludes the use of nasal cannulas
* Pregnancy and lactation period
* Inability to cooperate with staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-14 (Estimated); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Inspiratory oxygen fraction (FiO2) in the hypopharynx | 5 minutes after the start of each combination of breathing pattern, device type, fraction of inspired oxygen and preset flow
  Inspiratory oxygen fraction (FiO2) in the hypopharynx during high flow oxygen therapy through nasal cannula and face mask, and standard oxygen therapy through non-rebreather face mask different physiological conditions
Expiratory oxygen fraction (FeO2) in the hypopharynx | 5 minutes after the start of each combination of breathing pattern, device type, fraction of inspired oxygen and preset flow
  Expiratory oxygen fraction (FeO2) in the hypopharynx during high flow oxygen therapy through nasal cannula and face mask, and standard oxygen therapy through non-rebreather face mask different physiological conditions
Expiratory fraction of carbon dioxide (FeCO2) in the hypopharynx | 5 minutes after the start of each combination of breathing pattern, device type, fraction of inspired oxygen and preset flow
  Expiratory fraction of carbon dioxide (FeCO2) in the hypopharynx during high flow oxygen therapy through nasal cannula and face mask, and standard oxygen therapy through non-rebreather face mask different physiological conditions

SECONDARY OUTCOMES:
Respiratory rate (RR) | 5 minutes after the start of each combination of breathing pattern, device type, fraction of inspired oxygen and preset flow
  Respiratory rate (RR)
Peripheral oxygen saturation (SpO2) | 5 minutes after the start of each combination of breathing pattern, device type, fraction of inspired oxygen and preset flow
  Peripheral oxygen saturation (SpO2) during different physiological conditions
The ratio of oxygen saturation by pulse oximetry/inspiratory oxygen fraction to respiratory rate (ROX-index) | 5 minutes after the start of each combination of breathing pattern, device type, fraction of inspired oxygen and preset flow
  The ratio of oxygen saturation by pulse oximetry/inspiratory oxygen fraction to respiratory rate (ROX-index) during different physiological conditions
Comfort | 5 minutes after the start of each combination of breathing pattern, device type, fraction of inspired oxygen and preset flow
  Visual-analog scale (VAS) for comfort evaluation (from 1 to 10, 1-full comfort, 10-full comfort)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey I Yaroshetskiy, MD, PhD, ScD, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (1):
- Sechenov University Clinic#4, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared upon reasonable request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication of the results for 10 years.
Access Criteria: All data will be shared upon reasonable request

REFERENCES:
- [Background] Perkins GD, Ji C, Connolly BA, Couper K, Lall R, Baillie JK, Bradley JM, Dark P, Dave C, De Soyza A, Dennis AV, Devrell A, Fairbairn S, Ghani H, Gorman EA, Green CA, Hart N, Hee SW, Kimbley Z, Madathil S, McGowan N, Messer B, Naisbitt J, Norman C, Parekh D, Parkin EM, Patel J, Regan SE, Ross C, Rostron AJ, Saim M, Simonds AK, Skilton E, Stallard N, Steiner M, Vancheeswaran R, Yeung J, McAuley DF; RECOVERY-RS Collaborators. Effect of Noninvasive Respiratory Strategies on Intubation or Mortality Among Patients With Acute Hypoxemic Respiratory Failure and COVID-19: The RECOVERY-RS Randomized Clinical Trial. JAMA. 2022 Feb 8;327(6):546-558. doi: 10.1001/jama.2022.0028. PMID 35072713
- [Background] Ospina-Tascon GA, Calderon-Tapia LE, Garcia AF, Zarama V, Gomez-Alvarez F, Alvarez-Saa T, Pardo-Otalvaro S, Bautista-Rincon DF, Vargas MP, Aldana-Diaz JL, Marulanda A, Gutierrez A, Varon J, Gomez M, Ochoa ME, Escobar E, Umana M, Diez J, Tobon GJ, Albornoz LL, Celemin Florez CA, Ruiz GO, Caceres EL, Reyes LF, Damiani LP, Cavalcanti AB; HiFLo-Covid Investigators. Effect of High-Flow Oxygen Therapy vs Conventional Oxygen Therapy on Invasive Mechanical Ventilation and Clinical Recovery in Patients With Severe COVID-19: A Randomized Clinical Trial. JAMA. 2021 Dec 7;326(21):2161-2171. doi: 10.1001/jama.2021.20714. PMID 34874419
- [Background] He Y, Zhuang X, Liu H, Ma W. Comparison of the efficacy and comfort of high-flow nasal cannula with different initial flow settings in patients with acute hypoxemic respiratory failure: a systematic review and network meta-analysis. J Intensive Care. 2023 May 10;11(1):18. doi: 10.1186/s40560-023-00667-2. PMID 37165464
- [Background] Grieco DL, Maggiore SM, Roca O, Spinelli E, Patel BK, Thille AW, Barbas CSV, de Acilu MG, Cutuli SL, Bongiovanni F, Amato M, Frat JP, Mauri T, Kress JP, Mancebo J, Antonelli M. Non-invasive ventilatory support and high-flow nasal oxygen as first-line treatment of acute hypoxemic respiratory failure and ARDS. Intensive Care Med. 2021 Aug;47(8):851-866. doi: 10.1007/s00134-021-06459-2. Epub 2021 Jul 7. PMID 34232336
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908